CLINICAL TRIAL: NCT02494817
Title: Development of a HIV Prevention Toolkit for At-risk HIV-negative Male Couples
Brief Title: HIV Prevention Toolkit for HIV-negative Male Couples
Acronym: MCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Daniel J Feaster, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20140561; R34MH102098 (NIH)
Record Dates: First submitted 2015-07-07; First posted 2015-07-10 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: HIV
Keywords: HIV prevention; Toolkit; Male couples; Sexual agreements

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Placebo Comparator): Couples assigned to the control group will be directed to the website that only has the following: 1) module about learning about effective HIV prevention strategies, 2) sexual health resource center, and 3) a link to download a corresponding smartphone app that will include the sexual health resource center.
  Interventions: Behavioral: Male Couples Agreement Project
- Intervention group (Active Comparator): Couples assigned to the intervention group will first as individuals view general video about purpose of study and how to use website functions; timeline activity about their relationship; select top values about their relationship; learn about effective HIV prevention strategies; learn about sexual agreements; select what items they want to have in their agreement; explore a learning module about testing and view the sexual health resource center. As a couple, they will log back into the website to view and compare timelines and relationship values; watch a video about communicating more effectively; negotiate and decide together what items they want to include in their agreement; explore the sexual health resource center and/or any other modules from when they were logged into the website as individuals; download a corresponding smartphone app that will include a copy of their newly created agreement and sexual health resource center.
  Interventions: Behavioral: Male Couples Agreement Project

INTERVENTIONS:
Behavioral: Male Couples Agreement Project — Couples assigned to the intervention group will first as individuals view general video about purpose of study and how to use website functions; timeline activity about their relationship; select top values about their relationship; learn about effective HIV prevention strategies; learn about sexual agreements; select what items they want to have in their agreement; explore a learning module about testing and view the sexual health resource center. As a couple, they will log back into the website to view and compare timelines and relationship values; watch a video about communicating more effectively; negotiate and decide together what items they want to include in their agreement; explore the sexual health resource center and/or any other modules from when they were logged into the website as individuals; download a corresponding smartphone app that will include a copy of their newly created agreement and sexual health resource center.

SUMMARY:
Though technology is integrated into the lives of our target population, use of any particular technology will depend on the content delivered, aesthetic appeal, and overall design. Based on the completion and analysis of data from Phase 1, the investigators were able to obtain feedback on HIV-negative male couples' attitudes toward the original content in the prevention toolkit modules. The research team, along with the web-developers, used this feedback to specifically tailor the content of the modules to fit the unique needs of the intervention's target population: at risk HIV-negative male couples. For Phase 2, the investigators conducted focus groups at each site to help identify strengths and potential areas for improvement of the prevention toolkit, which will be incorporated before piloting it in the intervention for Phase 3 of this project. After assessing the acceptability of the prevention toolkit, including the content of modules, aesthetic appeal, and overall design with HIV-negative male couples target population, the research team will pilot test whether the RCT with the prevention toolkit will help reduce HIV risk through formation and adherence to a sexual agreement, reduction in occurrences of condomless anal sex with casual sex partners, and increase testing behaviors among at-risk HIV-negative male couples. The interactive website, herein referred to as the "HIV prevention toolkit" will contain unique modules about sexual agreements and effective HIV prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

Eligible male couples:

1. are identified as two men (i.e., main partners) who had been in a sexual relationship together for > 6 months;
2. are at least 18 years of age;
3. are self-reported as being HIV-negative;
4. had been practicing CAS in their relationship for > 6 months;
5. report no recent history (< 1 year) of intimate partner violence (IPV) or coercion;
6. have had no current sexual agreement; and
7. own a smartphone and have an alternate method to access the Internet (e.g., computer).

Exclusion Criteria:

1. Interested participants, including both men of a male couple, who did not meet the inclusion criteria above will be excluded from participating in Phase 3 of this study.
2. Individuals who participated in Phase 1 or 2 will be were excluded from participating in Phase 3 of this study.
3. Adults who are unable to consent;
4. Individuals who are not yet adults;
5. Pregnant and non-pregnant women, and prisoners.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason W Mitchell, PhD, Principal Investigator — University of Miami
Locations (1):
- Clinical Research Building, Miami, Florida, United States

REFERENCES:
- [Derived] Mitchell JW, Lee JY, Wu Y, Sullivan PS, Stephenson R. Feasibility and Acceptability of an Electronic Health HIV Prevention Toolkit Intervention With Concordant HIV-Negative, Same-Sex Male Couples on Sexual Agreement Outcomes: Pilot Randomized Controlled Trial. JMIR Form Res. 2020 Feb 13;4(2):e16807. doi: 10.2196/16807. PMID 32044754

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Couples assigned to the intervention group will first, as individuals, view general video about purpose of study and how to use website functions; timeline activity about their relationship; select top values about their relationship; learn about effective HIV prevention strategies; learn about sexual agreements; select what items they want to have in their agreement; explore a learning module about testing and view the sexual health resource center. As a couple, they will log back into the website to view and compare timelines and relationship values; watch a video about communicating more effectively; negotiate and decide together what items they want to include in their agreement; explore the sexual health resource center and/or any other modules from when they were logged into the website as individuals; download a corresponding smartphone app that will include a copy of their newly created agreement and sexual health resource center.
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 162 (representing 81 couples) | 136 (representing 68 couples)
3 Month Assessment | 125 (represents 59 couples and 7 partnered men) | 92 (represents 44 couples and 4 partnered men)
6 Month Assessment | 115 (represents 52 couples and 11 partnered men) | 98 (represents 45 couples and 8 partnered men)
Completed | 107 (49 couples and 9 partnered men completed all 3 assessments (baseline, 3- and 6-month)) | 87 (41 couples and 5 partnered men completed all 3 assessments (baseline, 3- and 6-month))
Not Completed | 55 | 49

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 162 | 136 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.55 (7.03) | 28.13 (7.33) | 27.81 (7.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 162 | 136 | 298
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 24 | 48
  Not Hispanic or Latino | 138 | 112 | 250
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 6 | 6
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 6 | 6 | 12
  White | 147 | 119 | 266
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 162 | 136 | 298
Sexual orientation [Count of Participants; unit: Participants]
  gay | 156 | 133 | 289
  bisexual | 6 | 3 | 9
Region of residence [Count of Participants; unit: Participants]
  Northeast | 19 | 11 | 30
  Midwest | 35 | 48 | 83
  South | 67 | 39 | 106
  West | 39 | 36 | 75
  US territory | 2 | 2 | 4
Education [Count of Participants; unit: Participants]
  Some High School | 7 | 3 | 10
  High School graduate / GED | 20 | 22 | 42
  Some college / AA / trade | 61 | 56 | 117
  Bachelors degree | 45 | 29 | 74
  Some grad school | 13 | 7 | 20
  Graduate degree | 14 | 19 | 33
  missing data | 2 | 0 | 2
Employment [Count of Participants; unit: Participants]
  Full time | 106 | 90 | 196
  Part time | 18 | 16 | 34
  Unemployed | 8 | 7 | 15
  On disability | 8 | 4 | 12
  Retired | 1 | 0 | 1
  Student | 21 | 19 | 40
Length of current relationship [Count of Participants; unit: Participants]
  3-6 months | 7 | 8 | 15
  6-12 months | 40 | 25 | 65
  1-3 years | 69 | 42 | 111
  3-6 years | 34 | 37 | 71
  6-10 years | 8 | 16 | 24
  10 + years | 4 | 8 | 12
Relationship status [Count of Participants; unit: Participants]
  Domestic partnership | 42 | 28 | 70
  Married | 24 | 40 | 64
  Engaged | 27 | 28 | 55
  None of the above | 62 | 31 | 93
  Other | 7 | 9 | 16
Relationship type [Count of Participants; unit: Participants]
  Monogamous | 153 | 117 | 270
  Open | 5 | 14 | 19
  No label and other | 3 | 5 | 8
  missing data | 1 | 0 | 1
Had sex with casual male partner (outside relationship) [Count of Participants; unit: Participants]
  Yes within last 3 months | 29 | 38 | 67
  No, not within last 3 months | 133 | 98 | 231
HIV testing frequency (before relationship) [Count of Participants; unit: Participants]
  Every 3-4 months | 24 | 15 | 39
  Every 6 months | 33 | 28 | 61
  Once a year | 29 | 30 | 59
  When I felt at risk for HIV | 19 | 18 | 37
  When I dated someone new | 6 | 4 | 10
  No testing pattern | 23 | 21 | 44
  Missing data | 28 | 20 | 48
HIV testing frequency (since in relationship) [Count of Participants; unit: Participants]
  Every 3-4 months | 8 | 0 | 8
  Every 6 months | 14 | 11 | 25
  Once a year | 26 | 23 | 49
  When I felt at risk for HIV | 16 | 20 | 36
  No testing pattern | 38 | 41 | 79
  Missing data | 60 | 41 | 101
When started having anal sex in relationship [Mean (Standard Deviation); unit: weeks] | 5.24 (10.25) | 5.96 (9.59) | 5.57 (9.95)
When started having condomless anal sex in relationship [Mean (Standard Deviation); unit: weeks] | 10.98 (20.09) | 22.91 (44.38) | 16.42 (31.18)

OUTCOME MEASURES:

1. Primary Outcome: Formation of a Sexual Agreement at 6 Months
Description: Self-reports of yes/no to forming a sexual agreement via electronic survey
Time Frame: 6 month
Population: For control, 115 men (52 dyads both partners provided data and 11 "dyads" where only one partner provided data) provided outcome data.
  For intervention, 98 men (45 dyads where both partners provided data and 8 "dyads" where only one partner provided data) provided outcome data.
  Only dyads where both partners provided data were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 104 | 90
Participants
  Formed an agreement | 56 | 66
  Did not form an agreement | 48 | 24

2. Primary Outcome: Adherence to a Sexual Agreement at 6 Months
Description: Self-report of yes/no of adhering to a sexual agreement
Time Frame: 6 month
Population: Participants who provided data in outcome 1 as having a concordant agreement were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 56 | 66
Participants
  Adhered to the agreement | 48 | 60
  Did not adhere to the agreement | 8 | 6

3. Secondary Outcome: Formation of a Sexual Agreement at 3 Months
Description: Self-reports of yes/no to forming a sexual agreement via electronic survey
Time Frame: 3 month
Population: 206 partnered men represent 44 dyads in the intervention arm and 59 dyads in the control arm, respectively. Couple-level findings are reported at the individual level.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 118 | 88
Participants
  Formed an agreement | 70 | 58
  Did not form an agreement | 48 | 30

4. Secondary Outcome: Adherence to a Sexual Agreement
Description: Self-reports of yes/no to adhering to a sexual agreement via electronic survey
Time Frame: 3 month
Population: Participants who provided data in outcome 3 as having a concordant agreement were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 70 | 58
Participants
  Adhered to the agreement | 62 | 54
  Did not adhere to the agreement | 8 | 4

5. Secondary Outcome: Had Condomless Anal Sex With Casual Male Sex Partner During Months 0-3
Description: Self-reports of yes/no of any anal sex with casual male sex partner between months and month 3 via electronic survey
Time Frame: 3 month
Population: 9 of 125 participants in control did not provide data, and 9 of 92 participants in intervention did not provide data.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 116 | 83
Participants
  Had CAS | 7 | 5
  Did not have CAS | 109 | 78

6. Secondary Outcome: Had Condomless Anal Sex With Casual Male Sex Partner Reported at Month 6
Description: Self-reports of yes/no any anal sex with casual male sex partner, measured at month 6 via electronic survey (about the previous 3 months, i.e., timeframe between months 3-6).
Time Frame: month 6
Population: Of control participants, only 104 of 115 provided data for this outcome. Of intervention participants, only 90 of 98 provided data for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 104 | 90
Participants
  Had CAS | 5 | 4
  Did not have CAS | 99 | 86

7. Secondary Outcome: Test for HIV During Past 3 Months (Months 0-3)
Description: Self-reports of yes/no via electronic survey taken at 3 month.
Time Frame: 3 month
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 125 | 92
Participants
  Yes, within last 3 months | 27 | 15
  No, not within last 3 months | 98 | 77

8. Secondary Outcome: Test for HIV During the Last 3 Months (Months 3-6)
Description: Self-reports of yes/no any test for HIV at month 6 assessment, collected via electronic survey for timeframe between months 3 and 6.
Time Frame: month 6
Population: 213 partnered men who completed 6-month assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 115 | 98
Participants
  Yes, within last 3 months | 27 | 11
  No, not within last 3 months | 88 | 87

ADVERSE EVENTS:
Time Frame: 6-months from baseline
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/162 | 0/136
Serious Adverse Events (participants affected / at risk) | 0/162 | 0/136
Other Adverse Events (participants affected / at risk) | 0/162 | 0/136

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Informed Consent Form (2015-06-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT02494817/ICF_000.pdf